CLINICAL TRIAL: NCT06957145
Title: Vista Protein Expression of Monocyte and T Cell Subsets in Multiple Sclerosis and Its Clinical Correlation: A 1-Year Follow-up Study
Brief Title: Vista Protein Expression of Monocyte and T Cell Subsets in Multiple Sclerosis and Its Clinical Correlation
Status: Recruiting | Type: Observational
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Rabia Gökcen Gozubatik Celik, Assoc. Prof., Koç University
Other Study IDs: Vista Protein Expression in MS
Record Dates: First submitted 2025-03-17; First posted 2025-05-04 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis, MS
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- People with MS: 30 People with MS
- Health Control: 30 Health Control

SUMMARY:
The aim of this study is to investigate whether VISTA, a newly identified negative immune regulatory protein, differs in monocytes and T cells of patients diagnosed with Multiple Sclerosis (MS) and Clinically Isolated Syndrome (CIS) compared to the same cell types in healthy controls. Additionally, the potential clinical correlation of VISTA expression in the follow-up of MS and CIS patients will be examined. By elucidating the role of VISTA in the pathophysiology of MS, this study will contribute to the literature by exploring its potential as a biomarker and its relevance in the development of novel therapeutic strategies.

Specifically, this study will compare VISTA protein secretion in MS patients at the time of their first attack with that of healthy controls. Furthermore, changes in VISTA protein secretion will be assessed in blood samples collected at 6- and 12-month follow-ups, and the correlations of these changes with clinical and laboratory findings will be investigated.

Finally, this study aims to determine whether CD4+ and CD8+ T cells, monocytes, and T regulatory (Treg) subgroups in the first attack blood samples of MS patients exhibit similar functional properties in terms of VISTA protein secretion as their counterparts in healthy controls. To achieve this, monocytes and T cell subtypes will be stimulated, and their pro- and anti-inflammatory cytokine responses will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older diagnosed with MS or CIS according to the 2017 McDonald criteria.
* No diagnosis of any autoimmune disease or malignancy.
* No new diagnosis of autoimmune disease or malignancy during the 1-year follow-up period.
* No use of antibiotics, nonsteroidal anti-inflammatory drugs (NSAIDs), or steroid treatments within one month prior to blood sampling.
* No vaccination within one month prior to blood sampling.
* Not in the menstrual cycle at the time of blood sampling.

Exclusion Criteria:

* Age below 18 years.
* Presence of a previous or newly diagnosed autoimmune disease or malignancy at the time of blood sampling.
* Use of antibiotics, nonsteroidal anti-inflammatory drugs (NSAIDs), or steroid treatments within one month prior to blood sampling.
* Vaccination within one month prior to blood sampling
* Being in the menstrual cycle at the time of blood sampling
* Patients without a definitive MS diagnosis according to the 2017 McDonald criteria will not be included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Multiple Sclerosis
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-06-30 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
VISTA Protein Secretion | Baseline, Week 0
  Comparison of VISTA protein secretion levels in blood samples of MS patients at the time of their first attack with those of healthy controls.

SECONDARY OUTCOMES:
Functional Comparison of Immune Cell Subsets via Cytokine Profiling and VISTA Expression Analysis | Baseline, Week 0
  VISTA protein expression levels in CD4+ and CD8+ T cells, monocytes, and regulatory T (Treg) cell subgroups from first attack blood samples of pwMS and healthy controls, measured by flow cytometry. VISTA protein secretion levels in the same cell subgroups, measured by multiplex cytokine assays. Cytokine responses (pro- and anti-inflammatory) in stimulated monocytes and T cell subsets, measured by flow cytometry and multiplex cytokine assays.
Clinical and Radiological Correlation | Baseline, Month 6, Month 12
  Demographic data, routine neurological examination findings, EDSS scores, cerebrospinal fluid (CSF) results, and MRI findings collected during the 1-year follow-up. Visual Evoked Potential (VEP) measurements during the same period. VISTA protein secretion levels and temporal changes measured by multiplex cytokine assays

CONTACTS AND LOCATIONS:
Overall Officials: Rabia G Gozubatik Celik, Assoc. Prof., Principal Investigator — Koç University
Locations (2):
- Turkey (Türkiye) (2):
  - Koc University, Istanbul, Istanbul
  - Bakirkoy Prof. Dr. Mazhar Osman Training and Research Hospital for Psychiatric, Neurologic and Neurosurgical Diseases, University of Health Sciences, Istanbul, Turkey, Istanbul

IPD SHARING:
Plan to Share IPD: No